CLINICAL TRIAL: NCT04318847
Title: Efficacy and Safety of the Administration of Ondansetron Versus Habitual Clinical Practice for the Treatment of Vomiting in Children With Mild and Moderate Dehydration: Randomized Clinical Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lizar Aguirre Pascasio (Other Government)
Responsible Party: Sponsor-Investigator, Lizar Aguirre Pascasio, Doctor in Medicine, Basque Health Service
Organization: Basque Health Service (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OND-URG
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Vomiting in Infants and/or Children
MeSH Terms: interventions — Ondansetron

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ondransetron (Experimental): Administration of ondansetron
  Interventions: Drug: Ondansetron 4 MG
- Habitual Clinical Practice (No Intervention): Habitual Clinical Practice

INTERVENTIONS:
Drug: Ondansetron 4 MG — Administration of ondansetron 4 mg or 8 mg according to weight
  Arms: Ondransetron

SUMMARY:
This clinical trial is intended to evaluate the efficacy and safety of the administration of ondansetron in children with mild-moderate dehydration.

The target population will be children between 4 and 13 years old who present vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least 2 vomits in the last 4 hours.
* Negative tolerance test.
* Signature of the informed consent by the parents or legal guardians.
* Diagnosis of vomiting or diagnosis of acute gastroenteritis with vomiting.
* Patients weighing 15 kg or more.

Exclusion Criteria:

* Altered conciousness.
* Sospected acute abdomen (appendicitis, invaginations...).
* Suspicion or presence of obstructive disease.
* Known severe digestive disease (Chron´s disease, ulcerative colitis...).
* Suspected food poisoning.
* Allergy to any of the drugs used in the study.
* Severe dehydration.
* Bilious vomiting.
* Previous abdominal surgery.
* Pathology that may affective degree of hydration of the patient (kidney failure, hypoalbuminemia..).
* Admission requirement or intravenous rehydration for any reason.
* Concomitant use of apomorphine.
* In relation to the possible lengthening of the QT, patients with problems of previous arrhythmia should be excluded or that they are receiving concomitant medication that can lengthen the QT, that have electrolyte disturbances.
* Patients receiving other serotonergic drugs.
* Patients who have undergone a previous adenotonsillectomy.
* Patients with hypocalcemia and/or hypomagnesemia.
* Patients with hereditary fructose intolerance.
* Diabetes patients.
* Lactose intolerant patients.
* Patients with indication of the low sodium diets.
* Hypersensitivity to ondansetron or other antagonists of the 5-HT3.

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Estimated)
Dates: Start 2021-10-10 (Estimated); Primary Completion 2023-04-10 (Estimated); Study Completion 2023-04-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of children who return to medical/pediatric consultation for de same episode | An average of 24 months
  Is calculated percentage of children who return to medical/pediatric consultation for de same episode of vomiting